CLINICAL TRIAL: NCT06378840
Title: An Exploratory Analysis of the Predictive Value of Immune Cell Using Single-cell Sequencing on the Outcome of Locally Advanced Cervical Cancer Treated by Concurrent Chemoradiotherapy Followed by PD-1 Inhibitor
Brief Title: the Predictive Value of Immune Cell in Locally Advanced Cervical Cancer
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2021-268-B
Record Dates: First submitted 2024-04-10; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Cervical Carcinoma; Concurrent Chemoradiotherapy; Immunotherapy
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Platinum; sintilimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue and blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: Nab-paclitaxel/Platinum, Sintilimab — Sintilimab Combined With Concurrent Nab-paclitaxel/Platinum-based Chemoradiotherapy

SUMMARY:
To explore the predictive value of immune cells by single-cell sequencing on the outcome of locally advanced cervical cancer treated by concurrent chemoradiotherapy Followed by PD-1 inhibitor

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the standard treatment for patients with locally advanced cervical cancer, but the treatment failure rate is up to 40% in previous studies. Immunotherapy using PD-1 inhibitor showed an objective response rate of 12-50% in studies, and pembrolizumab was approved by the US Food and Drug Administration for patients with advanced PD-L1-positive cervical cancer who experienced progression during or after chemotherapy. And according to KEYNOTE-A18, the addition of PD-1 inhibitor Pembrolizumab to the current concurrent chemoradiotherapy improved the PFS of such group of patients. But the detailed change of immune cells (tumor microenvironment and PBMC) during treatment is unknown, and studies on the relationship between immune cells and treatment-related side effect and efficiency is also in need.

ELIGIBILITY:
Inclusion criteria:

1. Age between 18 and 75;
2. Untreated patients with pathologically proven locally advanced cervical cancer;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
4. Adequate hematological, renal and hepatic functions:

   4.1 Hemoglobin > 8.0 g/dl 4.2 Neutrophils > 2000 cells/μl; Leukocytes > 4 × 109/L 4.3 Platelets > 100 × 109/Lg. 4.4 Serum urea nitrogen (BUN) ≤ 1.5 × upper normal limit (UNL) 4.5 Serum creatinine (Cr) ≤ 1.5 × upper normal limit (UNL) 4.6 Serum ALT/AST ≤ 2.5× UNL 4.7 Serum Total bilirubin ≤ 1.5× UNL
5. Life expectancy > 6 months
6. Eligible for concurrent chemoradiotherapy assessed by principle investigator;
7. No obvious active bleeding;
8. Written informed consent must be available before study registration

Exclusion criteria:

1. Recurrent or distant metastatic disease;
2. Prior malignancies (other than curable non-melanoma skin cancer) within 5 years;
3. Active autoimmune diseases requiring systemic treatment or other diseases requiring long-term use of substantial amount of hormones or other immunosuppressants;
4. Patients who need to receive systemic corticosteroids (dose equivalent to or higher than prednisone 10mg qd) or other immunosuppressants within 14 days before enrollment or during the study;
5. Vaccination of live attenuated vaccine 30 days before enrollment, or planned vaccination of live attenuated vaccine during the study;
6. Previous organ transplantation or HIV patients;
7. Allergic to macromolecular proteins /monoclonal antibodies, or to any test drug component;
8. Active acute or chronic viral hepatitis B or C. Hepatitis B virus (HBV) DNA> 2000IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA> 103 copies/ml.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced cervical carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the change of immune cells in the blood after chemoradiotherapy and immunotherapy | 1 year
  through single-cell sequence and data analysis, the investigators will focus on the percentage of each sub-type of immune cells after treatment, differential gene expression profiles in special cell type after chemoradiotherapy and immunotherapy.
the predictive value of the changed immune cell subtype in the blood on the side effect of immunotherapy | 1 year
  the investigators will focus on the occurrence and grade of side effect from immunotherapy according to the NCCN clinical practice guidelines in the evaluation and management of immunotherapy-related toxicity (through the symptoms, physical examination, and also through blood/image/endoscopy examination, such as blood routine, liver and renal function, TSH/T3/T4/ACTH concentration, myocardial enzymes concentration, EKG, echocardiography, CT/MRI, et al). And through statistical analysis, the investigators try to figure out if there is any immune subtype or any special molecular to a possible biomarker of the occurrence of any immunotherapy-related side effect.
the predictive value of the changed immune cell subtype in the blood on the effect of chemoradiotherapy and immunotherapy | 2 years
  through statistical analysis, the investigators try to figure out if there is any immune subtype or any special molecular to a possible biomarker of disease control (disease progression or not accordingly to the RECIST criterion)

SECONDARY OUTCOMES:
the change of immune cells in the tissue after chemoradiotherapy | 1 year
  through single-cell sequence and data analysis, the investigators will focus on the percentage of each sub-type of immune cells in the tumor microenvironment and differential gene expression profiles in special cell type after chemoradiotherapy.
the predictive value of the changed immune cell subtype in the tissue on the effect of chemoradiotherapy and immunotherapy | 2 years
  through statistical analysis, the investigators try to figure out if there is any immune subtype or any special molecular in the tumor tissue to a possible biomarker of disease control (disease progression or not accordingly to the RECIST criterion)
the predictive value of the changed immune cell subtype in the tumor microenvironment on the side effect of immunotherapy | 1 year
  through statistical analysis, the investigators try to figure out if there is any immune subtype or any special molecular in the tumor tissue to a possible biomarker of the occurrence of any immunotherapy-related side effect.

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided